CLINICAL TRIAL: NCT06437288
Title: Real-World Study of Hematoporphyrin Injection-Based Photodynamic Therapy in Patients with Recurrent or Residual Superficial Esophageal Cancer
Brief Title: Hematoporphyrin Photodynamic Therapy for Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian-jun Li, Prefessor, Endoscopy Department Administrative Director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-183
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Cancer; Photodynamic Therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- photodynamic therapy (Experimental): Receive an intravenous infusion of hematoporphyrin injection at a dose of 3mg/kg over 60 minutes.
  Undergo 630nm laser irradiation 48-72 hours after the infusion.
  Interventions: Procedure: photodynamic therapy

INTERVENTIONS:
Procedure: photodynamic therapy — Receive an intravenous infusion of hematoporphyrin injection

SUMMARY:
The objective of the present clinical trial is to assess the efficacy of photodynamic therapy (PDT) employing hematoporphyrin injection in the management of recurrent or residual superficial esophageal carcinoma. The principal objective is to determine the capability of this therapeutic modality to elicit a complete response in the patient cohort under investigation.

The central research question that this study seeks to address is as follows:

What is the rate of complete response at day 28 following treatment with photodynamic therapy utilizing hematoporphyrin injection in patients suffering from recurrent or residual superficial esophageal cancer? This study is designed as a single-arm trial, devoid of a control or comparison group.

Eligible participants will meet the following criteria:

They will be adult patients, aged between 18 and 80 years, who have experienced recurrence or retention of superficial esophageal cancer subsequent to prior therapeutic interventions.

They will receive an intravenous administration of hematoporphyrin injection at a dosage of 3mg/kg over a duration of 60 minutes.

They will undergo irradiation with a 630nm laser, which will be administered 48-72 hours post-infusion.

Their response to treatment will be evaluated at day 28 post-therapy, with assessments encompassing complete response, progression-free survival, overall survival, swallowing functionality, quality of life, and the incidence of adverse events throughout the duration of the study

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18 and 80 years (inclusive of both 18 and 80 years), with no restrictions on gender.

  2.Patients with esophageal squamous cell carcinoma who have undergone prior treatment, including radiotherapy, chemotherapy, immunotherapy, or surgical intervention (esophagectomy or endoscopic esophageal cancer surgery), with pathological confirmation of recurrence or residual disease (at least of high-grade intraepithelial neoplasia or above).

  3.Patients with superficial esophageal cancer, where the primary lesion is located in the mucosal or submucosal layer, and the muscular layer is still intact, as indicated by ultrasound endoscopy and related examinations.

  4.Subjects capable of tolerating general anesthesia. 5.Absence of severe hematological, coagulation, cardiac, pulmonary, hepatic, renal, or immunological abnormalities.

  6.Voluntary consent to participate in the clinical trial after being fully informed about the purpose, process, potential risks, and benefits of the trial, including the subject's obligations.

Exclusion Criteria:

1. Known allergy to the study medication or related drugs.
2. Patients who have not recovered from the toxicities associated with prior radiotherapy or chemotherapy treatments.
3. Previous treatment with other photosensitizers that was ineffective, or subjects who have received a photosensitizer treatment within 12 months prior to enrollment.
4. Use of other photosensitizing medications within 4 weeks prior to administration, such as tetracycline antibiotics, sulfonamides, and phenothiazines.
5. Neutrophil count <1.5×10^9 /L, platelet count <100×10^9 /L, or hemoglobin <100 g/L.
6. Serum creatinine ≥3 times the upper limit of normal or creatinine clearance <60 ml/min/1.73m^2; ALT or AST >3 times the upper limit of normal; or in the case of liver metastasis, ALT or AST >5 times the upper limit of normal; serum bilirubin >3 times the upper limit of normal.
7. Presence of severe comorbid conditions, including serious heart disease, cerebrovascular disease, uncontrolled diabetes, and uncontrolled hypertension.
8. HIV, HCV, syphilis infection, or positive for both hepatitis B surface antigen and e antigen.
9. Active esophageal inflammation (especially visible active ulcers, hyperemia, necrosis, etc. under endoscopy) or clinically significant active infection symptoms.
10. Pregnant or lactating women, and sexually active subjects of childbearing potential (including males) who refuse to use appropriate contraceptive measures during the study.
11. Active bleeding or bleeding diathesis (abnormal coagulation mechanism).
12. Severe physical or mental illness that may affect treatment, assessment, or compliance with the study protocol.
13. Concurrent second primary tumor undergoing treatment.
14. Single lesion greater than 5cm in length.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-09-18 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
The complete response rate evaluated by endoscopic ultrasound (EUS) | 56 days after the treatment.
  The proportion of patients showing a complete disappearance of the tumor following the treatment, as assessed by EUS on day 56

SECONDARY OUTCOMES:
Progression free survival | 3 years
  Length of time during and after the treatment of a disease, in which a patient lives with the disease but it does not get worse.
Overall survival | 3 years
  length of time from the start of the treatment until the death of the patient, regardless of the cause.
Adverse events | 1 month after the treatment
  Adverse events of the treatment.
Quality of life evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30(EORTC QLQ-C30) | 0.5 year; 1 year; 3 year
  The Quality of life evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30(EORTC QLQ-C30) assesses cancer patients' quality of life with 30 items in functional and symptom scales scored 1-3, and a global health scale scored 1-7. Higher scores on functional/global health scales indicate better quality of life, while higher symptom scores mean worse outcomes. The scale's minimum and maximum scores vary by the number of items in each scale, with transformation to a 0-100 scale for standardization.
Stooler's dysphagia grading | 0.5 year; 1 year; 3 year
  Stooler's dysphagia grading, in its full title, is known as the Stooler's Dysphagia Scale. This scale is used to assess the severity of dysphagia, which is difficulty or discomfort in swallowing. The Stooler's scale categorizes dysphagia into five grades, ranging from Grade 0 to Grade 4, with higher grades indicating more severe dysphagia.
  Here is a breakdown of the Stooler's Dysphagia Scale:
  Grade 0: No difficulty in swallowing. Grade 1: Occasional difficulty in swallowing solids. Grade 2: Occasional difficulty in swallowing liquids and frequent difficulty with solids.
  Grade 3: Complete inability to swallow solids and frequent difficulty with liquids.
  Grade 4: Inability to swallow any oral intake. In this scale, a lower grade indicates a better outcome, as it signifies less difficulty in swallowing. Conversely, a higher grade indicates a worse outcome, with Grade 4 being the most severe, indicating the inability to swallow anything orally.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic Department of Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China